CLINICAL TRIAL: NCT04333758
Title: Outpatient and Home Advanced Rehabilitation Therapeutics Using Jintronix Virtual Reality Telerehabilitation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Kuah Wee Keong Christopher, Principal Occupational Therapist, Tan Tock Seng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHG DSRB 2016/00442
Record Dates: First submitted 2020-03-17; First posted 2020-04-03 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: Rehabilitation, Telerehabilitation, Virtual Reality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Prospective open label study.
Oversight: FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Jintronix Intervention (Experimental): 2 consecutive phases of intervention for all participants using Jintronix virtual reality telerehabilitation software.
  Phase 1 consisted of 9 (3/week for 3 weeks) 45-min/session clinic-based sessions conducted by study team therapist, with concurrent caregiver training.
  Phase 2 consisted of 20 (5/week for 4 weeks) 45min/session home-based sessions supervised by trained caregiver, with telemonitoring by study team therapist.
  Interventions: Device: Jintronix Virtual Reality Telerehabilitation System

INTERVENTIONS:
Device: Jintronix Virtual Reality Telerehabilitation System — System consists of an internet-based rehabilitation software linked to a Microsoft Kinect camera for motion detection.
  Study team therapist prescribed a list of guided exercises and therapeutic activities (games) for training of whole body, lower and upper extremities. These can be done in sitting or standing, depending on individual participant's capacity.
  Telemonitoring is done by study team therapist during each of the training day (Mondays-Fridays) of the home-based training phase. Training performance results are reviewed and training games are adjusted or changed to optimise home training.
  Other Names: Jintronix

SUMMARY:
The use of virtual reality technology in a telerehabilitation service is not well established in Singapore. This feasibility trial aims to evaluate the benefits of using Jintronix to deliver a clinic-to-home, caregiver-supervised and individualised exercise telerehabilitation program to complement outpatient services and improve clinical outcomes for post-stroke users.

DETAILED DESCRIPTION:
With the emphasis on improving population health, reducing the need for hospital care, and promoting self-management, it will be beneficial to make good use of current available technologies to complement centre-based therapy with cost effectiveness and efficiency.

One mode of such care delivery to a patient's home is through a telerehabilitation system that enables remote monitoring of patients' participation and performance in individualised home exercises. In addition, timely review and adjustments in the home programs to cater to progress or changes in patients' performance can be carried out by therapists remotely.

In the recent years, there has been an increased utilisation of virtual reality applications in physical rehabilitation for specific training objectives, such as, movement retraining, balance control and strength training. Virtual reality exercises when prescribed with defined training objectives and duration can potentially be valuable to increase patients' training intensity in the comfort of their own homes.

The majority of patients receiving outpatient and home based rehabilitation at Tan Tock Seng Hospital (TTSH) Rehabilitation Centre (RC) and Centre for Advanced Rehabilitation Therapeutics (CART) are patients who have had a stroke. Hence this group of outpatients that are at least 3 months post-stroke will be recruited for this trial. It is hypothesized that they will benefit from increased intensity of upper limb, balance and/or gait rehabilitation with Jintronix telerehabilitation system that facilitates them to further exercise at home and not just at the clinic.

The study is thus designed to evaluate the feasibility of a novel telerehabilitation service based on the Jintronix Virtual Reality Platform to complement existing outpatient therapy services of TTSH RC (including its outpatient service arm at CART).

ELIGIBILITY:
Inclusion Criteria:

* patients with motor deficits due to stroke as diagnosed by CT or MRI, who are attending outpatient rehabilitation services at Tan Tock Seng Hospital Rehabilitation Centre and Centre for Advanced Rehabilitation Therapeutics
* post stroke of at least 3 months with stable neurological status
* 21-75 years old
* able to perform at minimal level of assistance (i.e. carer provides only up to 25% of physical support) for sitting, standing and/or walking tasks
* has a primary caregiver that must be present in all trial sessions
* able to understand and participate in a 15 minutes Jintronix trial during screening

Exclusion Criteria:

* has seizure history
* has severe cognitive deficits, perceptual deficits, and/or emotional-behavioural issues
* has unstable medical conditions which may affect participation (e.g unresolved sepsis, postural hypotension, end stage renal failure) or anticipated life expectancy of <1 year due to malignancy or neurodegenerative disorder
* has pain score of >5
* is pregnant or breastfeeding
* has known poor cardiac ejection fraction (<30%) or lung function (FEV1<30%)
* has non-weight bearing status in either lower extremities
* has caregiver who is unable to meet competency requirements as assessed by study team

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wee Keong Christopher Kuah, MSc, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Centre for Advanced Rehabilitation Therapeutics, Tan Tock Seng Hospital, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- Jintronix Intervention: 2 consecutive phases of intervention for all participants using Jintronix virtual reality telerehabilitation software.
  Phase 1 consisted of 9 (3/week for 3 weeks) 45-min/session clinic-based sessions conducted by study team therapist, with concurrent caregiver training.
  Phase 2 consisted of 20 (5/week for 4 weeks) 45min/session home-based sessions supervised by trained caregiver, with telemonitoring by study team therapist.
  Jintronix Virtual Reality Telerehabilitation System: System consists of an internet-based rehabilitation software linked to a Microsoft Kinect camera for motion detection.
  Study team therapist prescribed a list of guided exercises and therapeutic activities (games) for training of whole body, lower and upper extremities. These can be done in sitting or standing, depending on individual participant's capacity.
  Telemonitoring is done by study team therapist during each of the training day (Mondays-Fridays) of the home-based training phase. Training performance results are reviewed and training games are adjusted or changed to optimise home training.
Period: Overall Study
Arm/Group | Jintronix Intervention
Started | 35
Completed | 32
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There are 3 drop-outs from the study.
  years | 55.03 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There are 3 drop-outs from the study.
  Participants
    Female | 11
    Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: There are 3 drop-outs from the study.
  Participants
    Chinese | 27
    Malay | 2
    Indian | 1
    Others | 2
Region of Enrollment [Count of Participants; unit: Participants] — Population: There are 3 drop-outs from the study.
  Participants
    Singapore | 32
Handedness [Count of Participants; unit: Participants] — Population: There are 3 drop-outs from the study.
  Participants
    Right | 30
    Left | 2
Education, Customized [Count of Participants; unit: Participants] — Population: There are 3 drop-outs from the study.
  Participants
    Primary School | 5
    Secondary School | 2
    Institute of Technical Education | 3
    Polytechnic Education | 5
    Tertiary Education | 17
Gaming Experience: Yes, No [Count of Participants; unit: Participants] — Population: There are 3 drop-outs from the study.
  Participants
    Yes | 19
    No | 13
Post Stroke Duration, Continuous [Median (Inter-Quartile Range); unit: days] — Population: There are 3 drop-outs from the study.
  days | 320.50 [202.75 to 871.25]
Nature of Stroke: Infarct, Haemorrhage [Count of Participants; unit: Participants] — Population: There are 3 drop-outs from the study.
  Participants
    Infarct | 12
    Haemorrhage | 20
Side of Stroke: Left, Right, Bilateral [Count of Participants; unit: Participants] — Population: There are 3 drop-outs from the study.
  Participants
    Left | 16
    Right | 14
    Bilateral | 2
Involved Side: Left, Right [Count of Participants; unit: Participants] — Population: There are 3 drop-outs from the study.
  Participants
    Left | 14
    Right | 18

OUTCOME MEASURES:

1. Primary Outcome: Fugl Meyer Upper Limb Motor Assessment
Description: Measures motor impairment of upper limb recovery from a neurological insult. Range of scores from 0-66 points. Total score of 66 points with higher scores indicating better arm motor functions.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 36.52 (16.55)

2. Primary Outcome: Fugl Meyer Upper Limb Motor Assessment
Description: as for outcome 1
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 38.48 (16.55)

3. Primary Outcome: Fugl Meyer Upper Limb Motor Assessment
Description: as for outcome 1
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 39.17 (16.20)

4. Primary Outcome: Fugl Meyer Upper Limb Motor Assessment
Description: as for outcome 1
Time Frame: Week 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 40.00 (16.70)

5. Primary Outcome: Berg Balance Scale
Description: Measures static and dynamic balance abilities. Range of scores from 0-56 points. Total score of 56 points with higher scores indicating better balance functions.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 43.34 (9.99)

6. Primary Outcome: Berg Balance Scale
Description: as for outcome 5
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 47.17 (8.64)

7. Primary Outcome: Berg Balance Scale Score
Description: as for outcome 5
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 47.59 (9.53)

8. Primary Outcome: Berg Balance Scale
Description: as for outcome 5
Time Frame: Week 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 48.59 (8.97)

9. Primary Outcome: 6 Minute Walk Test
Description: Measures endurance inferred from distance measured directly via distance markers placed on ground, as the participant walked up and down repeatedly on a flat ground walking track for a duration of 6 minutes.
  Higher distance covered by participant in this 6 minutes indicates a better outcome of higher endurance. There is no lower and upper distance limits set for this measure.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
meters | 206.23 (129.38)

10. Primary Outcome: 6 Minute Walk Test
Description: as for outcome 9
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
meters | 227.67 (144.46)

11. Primary Outcome: 6 Minute Walk Test
Description: as for outcome 9
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
meters | 239.83 (148.56)

12. Primary Outcome: 6 Minute Walk Test
Description: as for outcome 9
Time Frame: Week 11
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
meters | 250.78 (158.95)

13. Primary Outcome: 10 Meter Walk Test
Description: Measures walking speed as participant walked on a flat ground walking track of 10 metres. Walking speed is calcuated by dividing 10 metres over time taken by a stopwatch.
  Faster walking speed indicates a better outcome. There is no lower and upper walking speed limits set for this measure.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
meters/second | 0.71 (0.42)

14. Primary Outcome: 10 Meter Walk Test
Description: as for outcome 13
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
meters/second | 0.74 (0.47)

15. Primary Outcome: 10 Meter Walk Test
Description: as for outcome 13
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
meters/second | 0.76 (0.51)

16. Primary Outcome: 10 Meter Walk Test
Description: as for outcome 13
Time Frame: Week 11
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
meters/second | 0.78 (0.52)

17. Primary Outcome: Numerical Pain Score
Description: Measures pain subjectively from participant's rating. Scale is from 0 (indicating no pain experienced) to 10 (indicating worst pain experienced).
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 0.10 (0.41)

18. Primary Outcome: Numerical Pain Score
Description: as for outcome 17
Time Frame: Week 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 0.103 [-0.112 to 0.319]

19. Primary Outcome: Numerical Pain Score
Description: as for outcome 17
Time Frame: Week 7
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 0.000 [0.000 to 0.000]

20. Primary Outcome: Numerical Pain Score
Description: as for outcome 17
Time Frame: Week 11
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | -0.103 [-0.397 to 0.190]

21. Primary Outcome: Stroke Self-Efficacy Questionnaire
Description: Measures a stroke survivor's perceived level of confidence in functional performance.
  Each of the 13 questions is scored on a 10-point scale (i.e. 0-10) with 0 indicating "Not At All Confident" and 10 indicating "Very Confident".
  The points from the 13 questions are then added to get a total score, with a minimum score of 0 and a maximum score of 130. Higher score reflects a better outcome.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 80.79 (19.30)

22. Primary Outcome: Stroke Self-Efficacy Questionnaire
Description: as for outcome 21
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 91.79 (20.11)

23. Primary Outcome: Stroke Self-Efficacy Questionnaire
Description: as for outcome 21
Time Frame: Week 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Jintronix Intervention
Number analyzed (Participants) | 32
score on a scale | 93.59 (20.49)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Jintronix Intervention
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

LIMITATIONS AND CAVEATS:
Results may be affected by participants having concurrent therapy, home exercise programs or other stroke-related treatment whilst undergoing the research, as these factors are not controlled for by this study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT04333758/Prot_SAP_000.pdf